CLINICAL TRIAL: NCT05702892
Title: Evaluation Of Biomarkers Associated With Bone Metabolism İn Patients With Different Periodontal Status
Brief Title: Evaluation of Bone Metabolism Biomarkers in Periodontal Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Ummuhan Tekin Atay, master in science, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ummuhan.tekinatay
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Periodontal Diseases
Keywords: periodontitis; saliva; sclerostin
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Sclerosteosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- periodontitis (Experimental)
  Interventions: Diagnostic Test: ELISA
- gingivitis (Experimental)
  Interventions: Diagnostic Test: ELISA
- periodontal healthy (Experimental)
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — ELISA(enzyme-linked immunosorbent assay)

SUMMARY:
This study evaluates the levels of biomarkers associated with bone metabolism in patients with different periodontal conditions.

DETAILED DESCRIPTION:
Background: In this study, the levels of bone metabolism markers found in the saliva of individuals with different periodontal conditions were compared and the relationship of these markers with periodontal status was examined.

Method: A total of 60 individuals, 20 with periodontitis (P), 20 with gingivitis (G), and 20 with periodontal healthy (S), were included in the study. Periodontal clinical parameters (plaque index, gingival index, bleeding on probing, clinical attachment level and probing pocket depth) and saliva samples were obtained from the individuals. Bone metabolism biomarker (necrotizing factor (TNF)-α, osteoprotegerin (OPG), nuclear factor kappa-β receptor activator ligand (RANKL) and sclerostin) levels in saliva samples were evaluated by enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old.
* not having any systemic disease that may affect periodontal status
* not smoking and alcohol use
* volunteer to participate in the study

Exclusion Criteria:

* periapical pathologies;
* resulting from orthodontics and occlusion extreme forces, including mechanical forces;
* chronic high-dose steroid therapy;
* radiation or immunosuppressive therapy;
* pregnancy;
* breastfeeding;
* allergy or sensitivity to any medication.
* Periodontal therapy or drug therapy for at least 6 months of study participants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of bone metabolism biomarkers in different periodontal conditions | baseline
  The levels of bone metabolism markers in the saliva of individuals with different periodontal status were compared and the relationship of these markers with periodontal status was examined.

SECONDARY OUTCOMES:
Probing pocket depth | baseline
  Probing pocket depth(PPD) was measured for determining the severity of the disease and clinical outcome. High probing depth shows more severe periodontal disease.
Gingival index | baseline
  The differences in gingival index scores between periodontally healthy and periodontitis.The gingival index was recorded for determining and classifying gingival status. The gingival index (Gİ) scores each site on a 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling and spontaneous bleeding.
Plaque index | baseline
  The differences in plaque index scores between periodontally healthy and periodontitis. Plaque index (PI) was recorded for determining and classifying oral hygiene status. The plaque index (PI) scores each site on a with 0 being no plaque in gingival area and 3 abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No